CLINICAL TRIAL: NCT02049814
Title: A Randomized, Open-label, Non-inferiority Study to Compare the Efficacy and Safety of Voglibose and Acarbose in Patients With Type 2 Diabetes Mellitus With Poor Control of Metformin
Brief Title: Efficacy and Safety of Voglibose Compared With Acarbose in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASCN1201; U1111-1147-3393 (Other: World Health Organization); VOG-P4-001 (Other: Takeda ID)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; voglibose; Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin + Voglibose 0.2 mg (Experimental): Metformin tablets, at the maximum tolerated dose ≥1000 mg/day, orally, for 12 weeks, in addition to voglibose 0.2 mg, tablets, orally, three times daily, for Weeks 1 and 2, followed by voglibose 0.3 mg, tablets, orally, three times daily, Weeks 3 through 12.
  Interventions: Drug: Metformin; Drug: Voglibose
- Metformin + Acarbose 50 mg (Active Comparator): Metformin tablets, at the maximum tolerated dose ≥1000 mg/day, orally, for 12 weeks, in addition to acarbose 50 mg, tablets, orally, three times daily, Weeks 1 and 2, then acarbose 100 mg, tablets, orally, three times daily, Weeks 3 through 12.
  Interventions: Drug: Metformin; Drug: Acarbose

INTERVENTIONS:
Drug: Metformin — Metformin tablets
  Other Names: Glucophage
Drug: Voglibose — Voglibose tablets
  Other Names: Basen
  Arms: Metformin + Voglibose 0.2 mg
Drug: Acarbose — Acarbose tablets
  Other Names: Glucobay, Precose, Prandase
  Arms: Metformin + Acarbose 50 mg

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of voglibose versus acarbose combined with metformin in participants with type 2 diabetes mellitus (T2DM) by evaluating levels of glycosylated hemoglobin.

DETAILED DESCRIPTION:
The drug being tested in this study is called voglibose. Voglibose is being tested to treat type 2 diabetes in people who have diabetes that is inadequately controlled on metformin alone. This study will look at glycemic control in people who take voglibose.

The study will enroll 494 patients. All participants will be enrolled in a 2-week screening phase and a metformin run-in phase. Eligible participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups:

* Metformin and Voglibose 0.2 mg
* Metformin and Acarbose 50 mg

All participants will be asked to take their current dose of metformin tablets and either voglibose or acarbose tablets three times a day throughout the study.

This multi-center trial will be conducted in China. The overall time to participate in this study is up to 20 weeks and participants will make 8 visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Has a historical diagnosis of type 2 diabetes mellitus (T2DM) for at least 6 months prior to the screening visit (V1).
2. Is male or female and aged from 18 to 75 years, inclusively.
3. Has a body mass index (BMI) between 20 and 45 kg/m^2, inclusively.
4. Is experiencing inadequate glycemic control with a glycosylated hemoglobin (HbA1c) concentration between 7.0% and 10.0%, inclusively.
5. Has been treated with Metformin for at least 3 months and at a stable dose (≥1000 mg/day) for at least 8 weeks prior to Screening, unless there is documentation that the participant's current dose is his or her maximum tolerated dose (MTD) and MTD is ≤1000 mg/day.
6. Keeps constant body weight with fluctuation range no more than 10% over for at least 3 months before screening.
7. Hemoglobin levels of the participant are ≥12 g/dL (≥120 g/L) in male and≥ 10 g/dL (≥100 g/L) in female at screening visit.
8. Male serum creatinine <1.5 mg/dL and female serum creatinine <1.4 mg/dL, or estimated glomerular filtration rate (eGFR) >60 ml/min/1.73m^2 based on calculation using the Modification of Diet in Renal Disease (MDRD) approximation at Screening.
9. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
10. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

1. Type 1 diabetes mellitus.
2. Has received insulin, voglibose, acarbose or other oral hypoglycemic drugs (except Metformin) for accumulative total of more than 7 days within the latest 3 months prior to Visit 1.
3. Has a history of cardiovascular disease: acute myocardial infarction, class III or IV heart failure, or cerebrovascular accident (stroke) within the latest 3 months prior to Visit 1.
4. The participant's liver function is damaged and has a significant clinical sign or symptom of hepatopathy, acute or chronic hepatitis, or the value of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is 3 times more than the upper limit of normal level at Visit 1.
5. Has an active proliferative retinopathy or macular degeneration that need to have an urgent treatment in the opinion of investigators.
6. Has a frequent attack of hypoglycemia or loses consciousness due to hypoglycemia in the opinion of investigators.
7. Has one or more times ketoacidosis or hyperosmotic status/coma.
8. Is receiving long-term (>14days) systemic glucocorticoid treatment (except the medicine: local, intraocular, inhalation or via the nose) or has received such treatment for 4 weeks at Visit 1.
9. Has a hematopathy (e.g. hemolytic anemia, drepanocytosis) that may interfere with the HbA1c test.
10. Has other liabilities (e.g. drug abuse, alcoholism or mental disorder) that may hinder the participant to follow and complete the study.
11. Has participated in another clinical study within the past 90 days or has received any investigational compound within 30 days prior to randomization.
12. Is unsuitable for this study in the opinion of investigators.
13. Has a disease need to use other taboo or caution drugs that is not listed in this study.
14. If female, is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2014-05-09 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (18):
- China (18):
  - Hefei, Anhui
  - Maanshan, Anhui
  - Beijing, Beijing Municipality
  - Guangzhou, Guangdong
  - Shenzhen, Guangdong
  - Taishan, Guangdong
  - Zhuzhou, Hunan
  - Nanjing, Jiangsu
  - Xuzhou, Jiangsu
  - Changchun, Jilin
  - Jilin, Jilin
  - Shenyang, Liaoning
  - Qingdao, Shandong
  - Shanghai, Shanghai Municipality
  - Yanan, Shanxi
  - Yan’an, Shanxi
  - Tianjin, Tianjin Municipality
  - Wenzhou, Zhejiang

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 22 investigative sites in China from 09 May 2014 to 28 June 2016.
Pre-assignment Details: Participants with a diagnosis of type 2 diabetes mellitus (T2DM) were enrolled in 1:1 to receive voglibose combined with metformin or acarbose combined with metformin.
Period: Overall Study
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg
Started | 248 | 246
Safety Set | 248 | 245
Completed | 219 | 219
Not Completed | 29 | 27
Not completed — Reason not Specified | 4 | 3
Not completed — Pregnancy | 1 | 0
Not completed — Lost to Follow-up | 2 | 3
Not completed — Serious Protocol Violation | 5 | 7
Not completed — Study Termination | 0 | 1
Not completed — Pretreatment event/Adverse Event (AE) | 8 | 5
Not completed — Voluntary withdrawal | 9 | 8

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included participants who took investigational product after randomization and had at least one efficacy assessment after treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg | Total
Number analyzed (Participants) | 236 | 233 | 469
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.41 (9.239) | 54.82 (9.386) | 54.62 (9.305)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 108 | 222
  Male | 122 | 125 | 247
Race/Ethnicity, Customized [Number; unit: participants]
  Ethnic Chinese | 236 | 233 | 469
Region of Enrollment [Number; unit: participants]
  China | 236 | 233 | 469
Height [Mean (Standard Deviation); unit: cm] | 164.8 (8.05) | 165.2 (8.07) | 165.0 (8.05)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.4 (3.27) | 26.4 (3.63) | 26.4 (3.45)
Baseline Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 126.2 (12.22) | 127.5 (12.69) | 126.8 (12.46)
Baseline Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 76.5 (7.69) | 77.7 (8.28) | 77.1 (8.00)
Baseline Pulse [Mean (Standard Deviation); unit: bpm] | 74.3 (7.73) | 75.4 (8.47) | 74.9 (8.12)
Baseline Temperature [Mean (Standard Deviation); unit: °C] | 36.3 (0.27) | 36.4 (0.25) | 36.3 (0.26)
Baseline Weight [Mean (Standard Deviation); unit: kg] | 71.6 (11.68) | 72.0 (12.09) | 71.8 (11.87)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 12
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 or final visit relative to baseline.
Time Frame: Baseline, Week 12
Population: Per Protocol Set (PPS) is a subset of FAS, including participants who completed treatment as was prescribed in protocol and had no important protocol deviation.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg
Number analyzed (Participants) | 156 | 156
percentage of glycated hemoglobin | -0.6982 (0.0742) | -0.9335 (0.0764)
Statistical Analysis 1: Comparison: Metformin + Voglibose 0.2 mg vs Metformin + Acarbose 50 mg; Test type: Non-Inferiority or Equivalence — If the upper limit of 95% CI of Least Square Mean (LS mean) of HbA1C Changes was less than 0.4%, it was considered that the non-inferiority was established; p = 0.0001, Paired t-test

2. Secondary Outcome: Change From Baseline in HbA1c at Week 6
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 6 relative to baseline.
Time Frame: Baseline and Week 6
Population: PPS is a subset of FAS, including participants who completed treatment as was prescribed in protocol and had no important protocol deviation.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg
Number analyzed (Participants) | 156 | 156
percentage of glycated hemoglobin | -0.4765 (0.0605) | -0.631 (0.0623)

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose Over Time
Description: The change between the fasting blood glucose value collected at weeks 6 and 12 or final visit relative to baseline.
Time Frame: Baseline, Weeks 6 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg
Number analyzed (Participants) | 156 | 156
mmol/L
  Change at Week 6 | -0.4234 (0.1397) | -0.8851 (0.1438)
  Change at Week 12 | -0.5041 (0.1398) | -0.8029 (0.1439)

4. Secondary Outcome: Change From Baseline in Postprandial Plasma Glucose (PPG) Over Time
Description: The change between the value of glucose after 1 and 2 hours of meal, measured by the meal tolerance test collected at Weeks 6 and 12 or relative to baseline.
Time Frame: 1 and 2 hours after meal at Baseline, Weeks 6 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg
Number analyzed (Participants) | 156 | 156
mmol/L
  Change at Week 6 (1 hour PPG) | -2.5149 (0.2308) | -3.8557 (0.2377)
  Change at Week 12 (1 hour PPG) | -2.1187 (0.2376) | -2.1187 (0.2376)
  Change at Week 6 (2 hour PPG) | -2.7461 (0.2553) | -4.0015 (0.2624)
  Change at Week 12 (2 hour PPG) | -2.6099 (0.2632) | -3.2347 (0.2705)

5. Secondary Outcome: Change From Baseline in Fasting Insulin at Week 12
Description: The change between the fasting insulin value collected at week 12 or final visit relative to baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: μU/dL
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg
Number analyzed (Participants) | 156 | 156
μU/dL | 0.0319 (1.1481) | 2.4169 (1.1959)

6. Secondary Outcome: Change From Baseline in Postprandial Serum Insulin at Week 12
Description: The change from Baseline in postprandial serum insulin, after 1 and 2 hours of meal collected at Week 12 relative to baseline.
Time Frame: 1 and 2 hours after meal at Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: μU/dL
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg
Number analyzed (Participants) | 156 | 156
μU/dL
  Change at Week 12 (1 hour) | -0.3435 (2.2504) | -1.44 (2.341)
  Change at Week 12 (2 hours) | 3.2972 (3.0059) | -0.1526 (3.1145)

7. Secondary Outcome: Change From Baseline in Fasting Glucagon at Week 12
Description: The change between the fasting glucagon value collected at week 12 or final visit relative to baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg
Number analyzed (Participants) | 156 | 156
pg/mL | 5.7543 (6.0009) | 11.4541 (6.2524)

8. Secondary Outcome: Change From Baseline in Postprandial Serum Glucagon at Week 12
Description: The change from Baseline in postprandial serum glucagon, after 1 and 2 hours of meal collected at Week 12 relative to baseline.
Time Frame: 1 and 2 hours after meal at Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg
Number analyzed (Participants) | 156 | 156
pg/mL
  Change at Week 12 (1 hour) | 20.4409 (5.683) | 15.69 (5.9068)
  Change at Week 12 (2 hours) | 34.8518 (6.41) | 13.0188 (6.6143)

9. Secondary Outcome: Change From Baseline in Calculated Homeostatic Model Assessment Insulin Resistance (HOMA IR) at Week 12
Description: The change between the value of HOMA-IR collected at Week 12 and HOMA-IR collected at Baseline. HOMA IR measures insulin resistance based on fasting glucose and insulin measurements: HOMA IR = fasting plasma insulin (µIU/mL) * fasting plasma glucose (mmol/L) / 22.5. A higher number indicates a greater insulin resistance.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Insulin resistance
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg
Number analyzed (Participants) | 156 | 156
Insulin resistance | -0.366 (0.5389) | 0.4983 (0.5596)

10. Secondary Outcome: Change From Baseline in Insulin Homeostatic Model Assessment Beta Cell Function (HOMA β) at Week 12
Description: The change between the value of HOMA-beta cell function collected at Week 12 and HOMA-beta cell function collected at Baseline. The homeostatic model assessment estimates steady state beta cell function as a percentage of a normal reference population (%B). HOMA %B = 20 * insulin (µIU/mL) / fasting plasma glucose (mmol/L) - 3.5.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage beta cell function
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg
Number analyzed (Participants) | 156 | 156
Percentage beta cell function | 15.3149 (5.4717) | 28.1739 (5.7253)

11. Secondary Outcome: Change From Baseline in Body Weight Over Time
Description: The change between body weight at weeks 2, 6 and 12 or relative to baseline.
Time Frame: Baseline, Weeks 2, 6 and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg
Number analyzed (Participants) | 156 | 156
kg
  Change at Week 2 | -0.016 (0.1661) | -0.1731 (0.1725)
  Change at Week 6 | -0.6315 (0.1412) | -0.7975 (0.1466)
  Change at Week 12 | -1.1563 (0.1878) | -1.4394 (0.1951)

ADVERSE EVENTS:
Time Frame: Up to Week 14
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety set included all randomized participants who received at least one dose of study treatment and had at least one subsequent safety assessment.
Arm/Group | Metformin + Voglibose 0.2 mg | Metformin + Acarbose 50 mg
Serious Adverse Events (participants affected / at risk) | 3/248 | 5/245
Other Adverse Events (participants affected / at risk) | 38/248 | 41/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin + Voglibose 0.2 mg (N=248) | Metformin + Acarbose 50 mg (N=245)
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
ALT increased (Investigations) | 0 | 1
Abnormal liver function test (Investigations) | 1 | 0
Cerebral ischemia (Nervous system disorders) | 1 | 0
Cerebral hemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Local swelling (General disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin + Voglibose 0.2 mg (N=248) | Metformin + Acarbose 50 mg (N=245)
Urinary tract infection (Infections and infestations) | 15 | 9
Flatulence (Gastrointestinal disorders) | 23 | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.